CLINICAL TRIAL: NCT06907979
Title: Experimental Manipulation of the Emotional Salience of Cannabis Use-Related Information in Regular Cannabis Users
Brief Title: Cannabis and Processing Emotions Study
Acronym: CAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Society of Addiction Psychology (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Samantha Fede, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00000423
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use Disorder, Severe
Keywords: cannabis; cannabis use disorder; emotional salience; problem recognition; problem awareness; transcranial magnetic stimulation; theta burst stimulation; TMS; TBS; medial orbitofrontal cortex; mOFC
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sham Theta Burst Stimulation (TBS) (Sham Comparator)
  Interventions: Device: TMS - Sham
- Intermittent Theta Burst Stimulation (iTBS) (Experimental)
  Interventions: Device: TMS - Active iTBS
- Continuous Theta Burst Stimulation (cTBS) (Experimental)
  Interventions: Device: TMS - Active cTBS

INTERVENTIONS:
Device: TMS - Sham — For sham TMS, participants will receive a placebo version of either cTBS or iTBS (in a counterbalanced order). To do this, we will use the "placebo" side of the TMS coil, which produces the same sound volume and sequence as active TMS but does not induce neuromodulatory effects due to using the opposite side of the TMS coil as the "active" side TMS coil. To simulate somatosensory effects of active TMS, sham TMS also use superficial stimulation with the same pulse sequence via a small electrode placed on the target region underneath the coil.
  Arms: Sham Theta Burst Stimulation (TBS)
Device: TMS - Active iTBS — Trains consisting of bursts of three stimuli at 50 Hz repeated at 5 Hz frequency delivered at 110% of measured individual motor threshold in 20 x 2-second trains with 8-second intertrain intervals (192 seconds total)
  Arms: Intermittent Theta Burst Stimulation (iTBS)
Device: TMS - Active cTBS — Trains consisting of bursts of three stimuli at 50 Hz repeated at 5 Hz frequency delivered at 110% of measured individual motor threshold in 1 x 40-second train (40 seconds total)
  Arms: Continuous Theta Burst Stimulation (cTBS)

SUMMARY:
The goal of this study is to test a causal neural mechanism of cannabis use-related problem recognition in individuals with severe cannabis use disorder using a non-invasive form of neuromodulation called transcranial magnetic stimulation (TMS). The main question it aims to answer is:

-Does manipulating neural activity in the medial orbitofrontal cortex of the brain affect cannabis use-related problem recognition?

Researchers will compare three forms of theta burst stimulation (TBS; sham, intermittent, and continuous) in each participant to see if manipulations in neural activity lead to changes in cannabis use-related problem recognition.

Participants will complete a screening interview about their mental health and substance use history and complete four in-person laboratory sessions, which involve questionnaires, four brief magnetic resonance imaging (MRI) scans, three TBS sessions, and three electroencephalogram (EEG) sessions. Participants will also be asked to provide urine samples and take saliva and/or breathalyzer tests at some of the lab visits.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for current, severe Cannabis Use Disorder (CUD), as assessed by the Structured Clinical Interview (SCID) for the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) during the screening interview
* Reports engagement in cannabis use at least four days per week, on average, over the past year
* Provide a urine sample positive for tetrahydrocannabinol (THC)
* Able to read and write in English
* Has used cannabis at least 20 days in the past month
* Endorses at least 10 distinct (of 40 possible) cannabis use-related problems across the screening interview and Lab Visit 1 questionnaires

Exclusion Criteria:

* Other non-cannabis illicit substance use more than once per month, on average, over the past year
* Current DSM-5 moderate or severe Alcohol Use Disorder, as assessed by the Structured Clinical Interview (SCID) for the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) during the screening interview
* History of bipolar I or psychosis spectrum disorders, as assessed by the SCID for DSM-5 during the screening interview
* Acute suicidality requiring treatment escalation, as assessed during the screening interview
* Currently taking any daily psychotropic medication
* Failure to meet standard MRI inclusion criteria (i.e., no presence of claustrophobia; cardiac pacemakers; neural pacemakers; surgical clips in the brain or blood vessels; surgically implanted metal plates, screws, or pins; cochlear implants; implanted uterine devices; metal braces; other metal objects in the body; history of significant injury to the brain or spinal cord; or pregnancy)
* Medical contraindications for transcranial magnetic stimulation (TMS; i.e., presence of a neurological disorder known to alter risk for seizures [e.g., stroke, aneurysm, brain surgery, structural brain lesion, brain injury, frequent/severe headaches], current medication therapy known to alter seizure threshold [e.g., clomipramine, Monoamine Oxidase inhibitors, imipramine, clozapine], recurrent seizures or epilepsy or family history of hereditary epilepsy, pregnancy, metallic implants in the body or other devices that may be affected by magnetic fields, or significant heart disease or cerebrovascular disease)
* History of allergies to cosmetics/lotions or EEG gel
* History of migraines
* Currently engaged in treatment for Cannabis Use Disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow (CBF) in the medial orbitofrontal cortex | Lab Visits 2 (day 8), 3 (day 15), and 4 (day 22)
  Function magnetic resonance imaging (fMRI) will be used to measure cerebral blood flow (CBF) in the medial orbitofrontal cortex (mOFC) using a 3-Tesla magnet. CBF values will be compared within-subject across stimulation conditions.
Amplitude of neurophysiological responses to self-referential cannabis use-related information | Lab Visits 2 (day 8), 3 (day 15), and 4 (day 22)
  Electroencephalogram (EEG) will be used to measure late positive potential (LPP) amplitudes to personalized auditory statements about cannabis-related positive expectancies and negative consequences, along with neutral stimuli. LPP amplitudes will be compared within-subject across stimulation conditions.

IPD SHARING:
Plan to Share IPD: Undecided